CLINICAL TRIAL: NCT00258115
Title: The Study of Inhibition of Inflammation in the Dysmetabolic Syndrome of Obesity
Brief Title: The Study of Inflammation on Blood Glucose Levels in Obese People
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CHS 03-48
Record Dates: First submitted 2005-11-22; First posted 2005-11-24 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Obesity
Keywords: Obesity; Metabolic Syndrome; Diabetes; Inflammation
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Diabetes Mellitus; Inflammation | interventions — salicylsalicylic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- salsalate (Active Comparator): 4.0 g/d divided dosing
  Interventions: Drug: salsalate
- placebo (Placebo Comparator): placebo for salsalate
  Interventions: Drug: salsalate

INTERVENTIONS:
Drug: salsalate

SUMMARY:
Chronic subaccute inflammation may underlie the development of diabetes cardiovascular disease and other components of the metabolic syndrome. Rodent studies suggest diet induced obesity is associated with activation of the IKK/NF-kB pathway and this pathway can be inhibited by salicylates. This study seeks to determine the effect of salicylates in overweight persons.

ELIGIBILITY:
Inclusion Criteria:

* obesity (> 85th% for age,BMI > 30); HbA1c <6%; hemoglobin and/or hematocrit within 2 standard deviations of normal range, without high risk of bleeding, without donation of blood in the previous 2 months; without involvement in any study evaluating an investigational drug or device for the previous 2 months; normal clotting studies; if female using barrier or oral contraception and with a negative pregnancy test.

Exclusion Criteria:

* Pregnant or lactating women; Patients with abnormal liver function defined as elevation of bilirubin, alkaline phosphatase, ALT, AST, or GGTP more than 1.5 times the upper limit of normal; Patients with kidney disease (serum creatinine > 1.5 mg/dL) macroalbuminuria (1+ protein on a standard urine dip-stick, or > 300 mg urinary albumin/day); (patients with microalbuminuria will be enrolled); Patients with any significant diseases or conditions, including emotional or psychiatric disorders and substance abuse, including history of binge drinking, that, in the opinion of the investigator, are likely to alter the patient's ability to complete the study ; Patients with metabolic acidosis (abnormal anion gap); History of gastric ulcer, dyspepsia, or upper or lower GI bleed; History of allergy to aspirin, or bleeding diathesis or currently on oral anticoagulants including warfarin, heparin, aspirin or other NSAIDs; Patients with major vascular event within 6 months of screening for the study (e.g., MI, stroke, CABG, angioplasty, PV surgery); Patients with chronic heart disease, or a history of myocardial infarction or stroke. Symptomatic angina pectoris or cardiac insufficiency as defined by the NYHA; classification as Functional Class III or IV; Patients who smoke more than one pack of cigarettes daily; Patients taking treatment medications known to affect insulin sensitivity (e.g. diuretics, beta-blockers); Patients with inadequately controlled serum lipid levels (total cholesterol ≥ 275 mg/dL and fasting triglycerides ≥ 450 mg/dL); Patients with history of cancer within 5 years prior to screening for the study other than basal cell carcinoma; active alcohol or other substance abuse.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2003-12; Primary Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
glycemia | one month

CONTACTS AND LOCATIONS:
Overall Officials: Allison B. Goldfine, MD, Principal Investigator — Investigator/Assistant Professor
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Shoelson SE, Lee J, Goldfine AB. Inflammation and insulin resistance. J Clin Invest. 2006 Jul;116(7):1793-801. doi: 10.1172/JCI29069. PMID 16823477
- [Background] Goldfine AB, Silver R, Aldhahi W, Cai D, Tatro E, Lee J, Shoelson SE. Use of salsalate to target inflammation in the treatment of insulin resistance and type 2 diabetes. Clin Transl Sci. 2008 May;1(1):36-43. doi: 10.1111/j.1752-8062.2008.00026.x. PMID 19337387
- [Result] Fleischman A, Shoelson SE, Bernier R, Goldfine AB. Salsalate improves glycemia and inflammatory parameters in obese young adults. Diabetes Care. 2008 Feb;31(2):289-94. doi: 10.2337/dc07-1338. Epub 2007 Oct 24. PMID 17959861
- See also: Joslin Diabetes Center Web-Site — http://www.joslin.org
- See also: Multicenter study to target inflammation using salsalate in type 2 diabetes. — http://tinsalt2d.org